CLINICAL TRIAL: NCT04682522
Title: Does the Microbiome Change With Flagyl Treatment After Ileocolic Resection for Crohn's Disease
Brief Title: Flagyl Microbiome in Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, sandykava, Surgeon, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20.1054
Record Dates: First submitted 2020-12-09; First posted 2020-12-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole (Active Comparator): Metronidazole 250 mg three times a day
  Interventions: Drug: Metronidazole Oral
- Standard care (No Intervention): Standard post-operative care, which may or may not include post-operative antibiotics

INTERVENTIONS:
Drug: Metronidazole Oral — 250 mg Three times a day
  Other Names: Flagyl
  Arms: Metronidazole

SUMMARY:
This study will compare the types of bacteria in the colon before and after colon resection surgery. The investigator will also compare standard post-operative antibiotic treatment to flagyl (metronidazole) treatment post-operatively to see if giving the antibiotic, decreases the incidence of return of Crohn's disease.

DETAILED DESCRIPTION:
Participants who are scheduled for colon resection for Crohn's disease will be invited to take part in this randomized study. Participants will be randomized 1:1 to either Metronidazole 250 mg three times a day, starting after surgery, for three months, or the local usual standard of care after surgery, which may be a different antibiotic prescribed by the physician.

Participants will also provide a stool sample at the following time points: prior to surgery, the day of discharge, at their follow-up appointment (usually about two weeks after surgery), three months, and six months.

Participants will also be followed to determine their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old who is deemed an acceptable surgical candidate for ileocolic resection.

Exclusion Criteria:

* any patients that are dependent on total parenteral nutrition and unable to tolerate oral intake
* patients who will undergo resection but will have an ileostomy created
* patients on maintenance antibiotics for their disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in bacteria in the gut | six months
  Any change in the types of bacteria in the gut during the study period. This will be done by doing genetic analysis of differences in stool over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Kavalukas, MD, Principal Investigator — University of Louisville
Locations (1):
- University Surgical Associates, Louisville, Kentucky, United States